CLINICAL TRIAL: NCT03681873
Title: Validation of an Extremely Low Dose Computed Tomography Protocol for Diagnosing Lung Nodules in Children and Young Adults
Brief Title: Validation of Low Dose CT for Diagnosis of Lung Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-6122
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Cancer; Metastasis to Lung
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Patients will receive both the clinically indicated and extremely low dose exams
  Interventions: Diagnostic Test: Extremely Low Dose CT

INTERVENTIONS:
Diagnostic Test: Extremely Low Dose CT — Patients undergoing a clinically indicated chest CT will also undergo the extremely low dose CT

SUMMARY:
The investigators have developed an extremely low dose computed tomography (CT) protocol that on preliminary testing has an effective dose in the range of two chest radiographs. The investigators plan to test this exam in patients with known or suspected cancer undergoing clinically indicated chest CT.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and young adult patients (ages 4 to <21 years)
* Known or suspected malignancy other than lymphoma
* Undergoing clinically indicated CT of the chest

Exclusion Criteria:

* Pregnancy identified by routine Department of Radiology verbal screening
* Prior enrollment in the same study (no patient will be enrolled more than once)
* Inability to provide consent and/or assent
* Lymphoma

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of extremely low dose CT | At time of imaging
  Sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center Burnet Campus, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thapaliya S, Gilligan LA, Brady SL, Anton CG, Crotty EJ, Nasser MP, Geller JI, Pressey JG, Zhang B, Dillman JR, Trout AT. Comparison of 0.3-mSv CT to Standard-Dose CT for Detection of Lung Nodules in Children and Young Adults With Cancer. AJR Am J Roentgenol. 2021 Dec;217(6):1444-1451. doi: 10.2214/AJR.21.26183. Epub 2021 Jul 7. PMID 34232694